CLINICAL TRIAL: NCT01388556
Title: PD4PD:Partnered Dance for Parkinson Disease
Acronym: PD4PD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Parkinson's Disease Foundation (Other)
Responsible Party: Principal Investigator, Gammon M. Earhart, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD4PD-09-0168; PDF (Other Grant/Funding Number: Parkinson's Disease Foundation)
Record Dates: First submitted 2011-06-29; First posted 2011-07-06 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson Disease
Keywords: exercise; Parkinson disease; motor symptoms; gait; balance
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tango (Experimental): Twice weekly tango dance classes for 12 months.
  Interventions: Behavioral: Tango dancing
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Tango dancing — Twice weekly tango dance classes
  Arms: Tango

SUMMARY:
Exercise is often noted as an important component in a comprehensive approach to the management of Parkinson disease (PD). Most studies of exercise have examined the effects of short-term interventions and have tested participants on their anti-Parkinson medications. As such, these studies have not been able to determine whether or not exercise may have a disease-modifying effect in people with PD. The investigators recent work has shown the potential benefits of dance as a form of exercise for individuals with PD, but, like previous work, has only examined short-term interventions. The investigators think that dance may be ideally suited for study over a longer period of time because dance incorporates many of the features recommended for inclusion in PD-specific exercise programs in a format that is known to be engaging and to enhance motivation to participate in healthful behaviors. As such, the investigators aim to determine both the short- and long-term effectiveness of a community-based dance program for individuals with Parkinson disease and to determine how physical function changes over time in individuals with PD who do not exercise as compared to those who exercise regularly. The investigators hypothesize that:

A) participation in dance will result in improved physical function, cognitive function, mood and quality of life in people with PD within 3 months,

B) additional improvements will be noted at 6 months as compared to 3 months,

C) improvements will be maintained at one year with continued, regular participation in a dance class,

D) those who do not exercise will show significant functional decline over a period of one year, a decline that will not be present in those who dance regularly.

ELIGIBILITY:
Inclusion Criteria:

* normal central and peripheral neurological function
* at least grade 4/5 strength and normal joint ranges of motion in both legs, - vision corrected to 20/40 or better
* able to walk independently for 10 feet with or without an assistive device, - normal somatosensory function in the feet (2-point discrimination, vibration, joint kinesthesia, and light touch)
* no history of vestibular disease

Exclusion Criteria:

* serious medical problem
* evidence of abnormality other than PD-related changes on brain imaging (previously done for clinical evaluations-not part of this research)
* history or evidence of neurological deficit other than PD that could interfere, such as previous stroke or muscle disease
* history or evidence of orthopedic, muscular, or psychological problem

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Motor Symptom Severity | 12 months
  We will use the Unified Parkinson Disease Rating Scale, Motor Subscale 3, to assess the severity of movement-related symptoms. This is a standanrdized and well-established tool composed of multiple items each scored on a 0-4 scale, with 0 indicating no impairment and 4 indication severe impairment. The overall severity of motor symptoms is determined by summing scores for all of the individual items.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Duncan RP, Earhart GM. Measuring participation in individuals with Parkinson disease: relationships with disease severity, quality of life, and mobility. Disabil Rehabil. 2011;33(15-16):1440-6. doi: 10.3109/09638288.2010.533245. Epub 2010 Nov 20. PMID 21091047
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886